CLINICAL TRIAL: NCT04923711
Title: A Perspective Randomized Controlled Study of the Formulation and Efficacy of Exercise Prescription for Patients With Coronary Heart Disease
Brief Title: Formulation and Efficacy of Exercise Prescription for Patients With Coronary Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jing Ma (Other)
Responsible Party: Sponsor-Investigator, Jing Ma, Clincial professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-249
Record Dates: First submitted 2021-05-31; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Coronary Heart Disease
Keywords: exercise prescription; cardiac rehabilitation; coronary heart disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity Group (Experimental): Group received a moderate exercise prescription of moderate intensity
  Interventions: Behavioral: Moderate intensity exercise prescription
- High Intensity Group (Experimental): Group received a moderate exercise prescription of high intensity
  Interventions: Behavioral: High intensity exercise prescription

INTERVENTIONS:
Behavioral: Moderate intensity exercise prescription — Exercise Intensity： Low-risk patients: the lower of 60-69% reserve heart rate or the heart rate at the anaerobic threshold.
  Moderate-risk or high-risk patients: the lower of 50-59% reserve heart rate or the heart rate at the anaerobic threshold.
  Arms: Moderate Intensity Group
Behavioral: High intensity exercise prescription — Exercise Intensity： Low-risk patients: the lower of 70-85% reserve heart rate or the heart rate at the anaerobic threshold.
  Moderate-risk or high-risk patients: the lower of 60-70% reserve heart rate or the heart rate at the anaerobic threshold.
  Arms: High Intensity Group

SUMMARY:
The purposes of this study is to standardize the process of formulating exercise prescriptions for coronary heart disease（CHD）, verify the safety and effectiveness of exercise prescriptions, and establish a database of exercise prescriptions for CHD, with a view to providing new solutions for cardiac rehabilitation.

DETAILED DESCRIPTION:
This study conducted a comparative study on the therapeutic effect and safety of exercise prescriptions for patients with coronary heart disease with different risk stratifications. The purposes of this study is to standardize the process of formulating exercise prescriptions for coronary heart disease（CHD）, verify the safety and effectiveness of exercise prescriptions, and establish a database of exercise prescriptions for CHD, with a view to providing new solutions for cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old with a diagnosis of coronary heart disease，NYHA class I-III HF patients.

Exclusion Criteria:

* acute myocardial infarction within 2 weeks
* Uncontrolled tachycardia (heart rate at rest >120bpm
* Uncontrolled polypnea（breath rate at rest >30 breath per minute
* Uncontrolled respiratory failure （SPO2 ≤90%）
* Uncontrolled hyperglycemia (Random blood glucose>18mmol/L)
* Uncontrolled malignant arrhythmia with hemodynamic instability
* Uncontrolled septic shock and septicopyemia
* Uncooperation of the patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of MACE | 6 month
  any incidence of the following: death, cardiac death, AMI, revascularization, stroke
The score of Seattle Angina Questionnaire increased | 6 month
  The score of Seattle Angina Questionnaire (SAQ, 0-100 each dimension, higher means greater condition）increased.
Routine color Doppler echocardiography changed. | 6 month
  Routine color Doppler echocardiography changed.
Improvement of Cardiopulmonary exercise test | 6 month
  the improvement of maximum oxygen uptake
Improvement of 6-minute walk test | 6 month
  the improvement of 6 minute walking distance
Improvement of grip strength test | 6 month
  the improvement of grip strength

SECONDARY OUTCOMES:
The score of Medical Outcomes Study Questionnaire Short Form 36 Health Survey (36-Item Short Form Survey) increased | 6 month
  The score of Medical Outcomes Study Questionnaire Short Form 36 Health Survey (abbreviation form is 36-Item Short Form Survey) increased. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability, The sections consists of Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, and Mental health. The total score of SF 36 Health survey is higher, the quality of life is higher.
The score of Patient Health Questionnaire decreased | 6 month
  The score of patient health questionnaire (PHQ9, normal range 0-27，indicating the profile of depression with the higher score) decreased
The score of Generalized Anxiexy Disorde-7 decreased | 6 month
  The score of Generalized Anxiexy Disorde-7 (GAD7, normal range 0-21，indicating the profile of anxiety with the higher score) decreased
The score of Chinese perceived stress scale decreased. | 6 month
  The score of Chinese perceived stress scale (CPSS, 0-56, higher means more stress) decreased.
The score of Pittsburgh Sleep Quality Index Scale decreased. | 6 month
  The score of Pittsburgh Sleep Quality Index Scale (PSQI, 0-21, higher means poorer sleep quality）decreased.
The score of Fagerstrom Test for Nicotine Dependence decreased. | 6 month
  The score of Fagerstrom Test for Nicotine Dependence (FTND, 0-10, higher means more dependence on nicotine）decreased.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ma, Principal Investigator — Department of Cardiology in Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: The IPD of the publication will be shared, including characteristic data, results, clinical follow up data.